CLINICAL TRIAL: NCT04192357
Title: A Randomised Controlled Trial of a Weight Loss Maintenance Program for Adults With Obesity: The WLM3P Study
Acronym: WLM3P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa (Unknown); CINTESIS@RISE, NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WLM3P01
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLM3P (Experimental): Participants will receive the M3F program. The M3F program is divided into three phases, being the first two of weight loss and the third phase of weight maintenance.
  Interventions: Behavioral: WLM3P
- Low-carb diet (Active Comparator): Participants will receive the low-carb diet program. The low-carb diet program is divided into two phases, being the first of weight loss which follows a low carb diet, and a second phase of weight maintenance.
  Interventions: Behavioral: Low-carb diet

INTERVENTIONS:
Behavioral: WLM3P — 18 months behavioral weight loss program divided into three phases (first and second phase of weight loss, during 1 month and 5 months, respectively; and a third phase of weight maintenance, during 12 months).
  Arms: WLM3P
Behavioral: Low-carb diet — 18 months behavioral weight loss program divided in two phases (first of weight loss during 6 months and a second phase of weight maintenance during 12 months).
  Arms: Low-carb diet

SUMMARY:
The aim of this study is to evaluate the effectiveness of a Weight Loss Maintenance 3 Phases Program (WLM3P) in maintaining long-term weight loss (at least 5% of initial body weight loss at 18 months), compared to a standard low carbohydrate diet (LCD) in adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years
* BMI ≥ 30 kg/m2 and ≤ 39.9 kg/m2
* Interested in being enrolled in a weight loss program
* Available to comply with study protocol and sign informed consent

Exclusion Criteria:

* Pregnant, breastfeeding or planning to become pregnant within the study period.
* Subjects with chronic inflammatory bowel disease (clinical history of Crohn's disease, ulcerative colitis, irritable colon and diverticulitis)
* Subjects with hormonal or thyroid pathology (hyper and hypothyroidism where TSH is not within normal range)
* Subjects with renal impairment
* Subjects with chronic liver disease other than non-alcoholic hepatic steatosis
* Subjects with autoimmune diseases and/or chronic use of corticosteroids.
* Use of weight loss medications/other nutritional supplements
* Subjects with psychiatric or neurological illness
* Subjects sensitive to any component of supplements
* Subjects with surgery or hospitalization in the last 30 days
* Subjects prescribed with 5 or more drugs
* Previous attempt to lose weight in the last month and/or weight loss of more than 10kg in the 3 months prior to the start of the study
* Subjects with excessive alcohol consumption (self-reported: drinking more than 3 glasses of wine/day - or equivalent)
* Subjects with history of drug, alcohol or other substances abuse.
* Eating behavior disorders
* Pacemaker carrier
* Urinary incontinence
* Vegetarians or vegans
* Subjects underwent bariatric surgery
* Type 1 or type 2 diabetes mellitus
* Altered blood clotting
* Severe heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 18 months
  Difference between the intervention and control group in the change of weight from baseline to the end of follow-up.

SECONDARY OUTCOMES:
Change in total fat mass | 18 months
  Difference between the intervention and control group in the change of total fat mass, measured by bioimpedance analysis from baseline to the end of follow-up.
Change in waist circumference | 18 months
  Difference between the intervention and control group in the change of waist circumference from baseline to the end of follow-up.
Change in body mass index | 18 months
  Change in body mass index (calculated as change in kg/m2, weight in kilograms, height in meters) from baseline to the end of follow-up.
Change in systolic and diastolic blood pressure | 18 months
  Difference between the intervention and control group in the change in systolic and diastolic blood pressure from baseline to the end of follow-up.
Change in intestinal microbiota | 18 months
  Difference between the intervention and control group in the change of intestinal microbiota from baseline to the end of follow-up.
  Bacterial DNA will be extracted from fecal samples. 16SRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Change in fasting plasma glucose concentrations | 18 months
  Difference between the intervention and control group in the change of serum glucose concentrations from baseline to the end of follow-up.
Change in fasting plasma insulin concentrations | 18 months
  Difference between the intervention and control group in the change of serum insulin concentrations from baseline to the end of follow-up.
Change in fasting plasma triglycerides concentrations | 18 months
  Difference between the intervention and control group in the change of serum triglycerides concentrations from baseline to the end of follow-up.
Change in fasting plasma low density lipoprotein (LDL) concentrations | 18 months
  Difference between the intervention and control group in the change of serum low density lipoprotein (LDL) concentrations from baseline to the end of follow-up.
Change in fasting plasma high density lipoprotein (HDL) concentrations | 18 months
  Difference between the intervention and control group in the change of serum high density lipoprotein (HDL) concentrations from baseline to the end of follow-up.
Change in fasting plasma glycated hemoglobin A1c (HbA1c) concentrations | 18 months
  Difference between the intervention and control group in the change of serum glycated hemoglobin A1c (HbA1c) concentrations from baseline to the end of follow-up.
Change in alanine aminotransferase (ALT) concentrations | 18 months
  Difference between the intervention and control group in the change of alanine aminotransferase (ALT) concentrations from baseline to the end of follow-up.
Change in aspartate aminotransferase (AST) concentrations | 18 months
  Difference between the intervention and control group in the change of aspartate aminotransferase (AST) concentrations from baseline to the end of follow-up.
Change in gamma-glutamyl transpeptidase (GGT) concentrations | 18 months
  Difference between the intervention and control group in the change of gamma-glutamyl transpeptidase (GGT) concentrations from baseline to the end of follow-up.
Change in HOMA-IR | 18 months
  Difference between the intervention and control group in HOMA-IR (homeostasis model assessment of insulin resistance) from baseline to the end of follow-up, calculated using the formula: fasting plasma glucose (mmol/L) x Fasting insulin (mIU/L)/22.5.
Change in creatinine concentrations | 18 months
  Difference between the intervention and control group in the change of creatinine concentrations from baseline to the end of follow-up.
Change in vitamin D concentrations | 18 months
  Difference between the intervention and control group in the change of vitamin D concentrations from baseline to the end of follow-up.
Change in high-sensitivity C-reactive protein (hs-CRP) concentrations | 18 months
  Difference between the intervention and control group in the change of high-sensitivity C-reactive protein (hs-CRP) concentrations from baseline to the end of follow-up.
Change in sodium concentrations | 18 months
  Difference between the intervention and control group in the change of sodium concentrations from baseline to the end of follow-up.
Change in potassium concentrations | 18 months
  Difference between the intervention and control group in the change of potassium concentrations from baseline to the end of follow-up.
Change in magnesium concentrations | 18 months
  Difference between the intervention and control group in the change of magnesium concentrations from baseline to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS, NOVA Medical School
Locations (1):
- NOVA Medical School, NOVA University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pereira V, Cuevas-Sierra A, de la O V, Salvado R, Barreiros-Mota I, Castela I, Camelo A, Brandao I, Santo CE, Faria A, Calhau C, Silvestre MP, Moreira-Rosario A. Gut Microbiota Shifts After a Weight Loss Program in Adults with Obesity: The WLM3P Study. Nutrients. 2025 Jul 18;17(14):2360. doi: 10.3390/nu17142360. PMID 40732984
- [Derived] Pereira V, Barreiros-Mota I, Cortez F, Castela I, Teixeira D, Calhau C, Camila Dias C, Moreira-Rosario A, Silvestre MP. A randomized controlled trial of a weight loss maintenance program in adults with obesity: the WLM3P study. Eur J Clin Nutr. 2024 Aug;78(8):694-702. doi: 10.1038/s41430-024-01454-4. Epub 2024 Jun 6. PMID 38844671